CLINICAL TRIAL: NCT00753480
Title: A Phase I, Open-Label, Dose-Escalation Study of the Safety and Pharmacokinetics of D4064A Administered Intravenously to Patients With Recurrent or Persistent Epithelial Ovarian, Primary Peritoneal, or Fallopian Tube Cancer After a Platinum-Containing Regimen
Brief Title: A Study of D4064A Administered to Patients With Recurrent or Persistent Epithelial Ovarian, Primary Peritoneal, or Fallopian Tube Cancer
Status: Suspended | Phase: Phase 1 | Type: Interventional
Sponsor: Genentech, Inc. (Industry)
Responsible Party: Clinical Trials Posting Group, Genentech, Inc.
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DMU4506g
Record Dates: First submitted 2008-09-12; First posted 2008-09-16 (Estimated); Last update posted 2008-11-07 (Estimated); Status verified 2008-11

CONDITIONS: Fallopian Tube Cancer; Ovarian Cancer; Peritoneal Cancer
Keywords: EOC; PPC; FTC
MeSH Terms: conditions — Fallopian Tube Neoplasms; Ovarian Neoplasms

INTERVENTIONS:
Drug: D4064A

SUMMARY:
This is a Phase I, multicenter, open-label, dose-escalation study of single-agent D4064A administered by IV infusion to patients with recurrent or persistent epithelial ovarian cancer (EOC), primary peritoneal cancer (PPC), and fallopian tube cancer (FTC) who have previously received a platinum-containing regimen. The study will enroll up to 56 patients at up to six investigative sites in the United States.

ELIGIBILITY:
Inclusion Criteria:

* ECOG performance status of 0 or 1
* Advanced, histologically documented epithelial ovarian, primary peritoneal, or fallopian tube cancer that has progressed or relapsed during or within 12 months of treatment with a platinum-containing chemotherapy regimen, and for which no standard therapy exists
* History of receiving five or fewer prior chemotherapy-containing regimens for EOC, PPC, or FTC (including primary therapy)

Exclusion Criteria:

* Prior treatment with chemotherapy or experimental anti-cancer agents within 4 weeks prior to Day 1
* Prior treatment with oregovomab (OvaRex(R)) or abagovomab
* History or clinical evidence of central nervous system or brain metastases
* Grade ≥ 2 peripheral neuropathy
* History of severe allergic or anaphylactic reactions to human, humanized, chimeric, or murine monoclonal antibodies
* History of clinically symptomatic liver disease, including viral or other hepatitis, history of or current alcoholism, or cirrhosis
* Untreated or persistent/recurrent malignancy (other than EOC, PPC, or FTC)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Estimated)
Dates: Start 2008-09

PRIMARY OUTCOMES:
Incidence and nature of dose-limiting toxicities (DLTs) | Length of study

SECONDARY OUTCOMES:
Incidence, nature, and severity of adverse events | Length of study
Incidence of anti-D4064A antibodies | Length of study
Changes in vital signs and clinical laboratory results | Length of study

CONTACTS AND LOCATIONS:
Overall Officials: Scott Holden, M.D., Study Director — Genentech, Inc.
Locations (2):
- United States (2):
  - Investigational Site, New York, New York
  - Investigational Site, Nashville, Tennessee